CLINICAL TRIAL: NCT02741505
Title: Open Masking, Micro Motionlogger Actigraph, 3T Siemens MRI, Sleep Deprivation, Nocturnal PSG
Brief Title: Brain Sleep Deprivation MRI Effects (BEDTIME)
Acronym: BEDTIME
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was not obtained
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-00971
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer's Disease
Keywords: cerebrospinal fluid (CSF); sleep; Obstructive Sleep Apnea (OSA); Sleep Disordered Breathing (SDB); Period Limb Movement during Sleep (PLMS)
MeSH Terms: conditions — Alzheimer Disease; Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Sleep Deprivation followed by Normal Sleep (Experimental): Subjects will be sleep deprived at the sleep laboratory.
  Interventions: Device: Actigraph

INTERVENTIONS:
Device: Actigraph — Participants will be asked to wear an actigraph

SUMMARY:
The primary purpose of this study is to explore the underlying mechanisms that link sleep to Alzheimer's disease (AD), with special focus on the clearance of metabolites in the extracellular space of the brain during sleep. Subjects will wear an actigraph for 1 week to determine regular daytime activity and sleep patterns. Subjects will then undergo partial sleep deprivation followed by 4 hours of in-lab nocturnal polysomnography (NPSG). Participants will be be asked to stay awake and active all day after the partial sleep deprivation with a new actigraphy secured by a hospital band to assure participants remain awake. They will seep inside an MRI machine for 90 minutes on the following night during their usual bedtime (established by 1 week actigraphy study.) Morphologic imaging, flow imaging and diffusion kurtosis imaging (DKI) will be performed on a 3T Siemens scanner.

ELIGIBILITY:
Inclusion Criteria:

* Age range 21-30
* Capable of giving informed consent

Exclusion Criteria:

* Diagnosis of any brain disease or brain damage including significant trauma, hydrocephalus, seizures, mental retardation or other serious neurological disorders (e.g. Parkinson's disease or other movement disorders). Persons with silent cortical infarcts will be excluded. White matter lesions will not be exclusions.
* History of major psychiatric illness (e.g., schizophrenia, bipolar or life long history of major depression)
* Conditions that alter normal sleep patterns: irregular sleep-wake rhythms (based on one week at home monitoring with actigraphy), moderate to severe periodic limb movement while you sleep (PLMS) or Obstructive Sleep Apnea (OSA).
* History of claustrophobia.
* BMI≥30
* Significant history of alcoholism or drug abuse.
* Inability to avoid the use of alcohol or caffeine during the 48h before the MRI.
* Current pregnancy or intent to become pregnant during the period of study.
* Any electronic or ferromagnetic devices (e.g., pacemaker or surgical clips) that constitutes a hazard for MRI imaging.
* Any medications adversely affecting cognition, blood pressure, glucose metabolism, or sleep will result in exclusion.

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Measure of Interstitial Space Volume during sleep using MRI imaging | 6 Months
  Data will be acquired using imaging sequences that comply with federal limits regarding radiofrequency energy deposition and gradient slew rates.

SECONDARY OUTCOMES:
Changes in Cerebral Spinal Fluid volume measured by increases in the power of slow wave activity (SWA) | 6 Months
  Data will be acquired using imaging sequences that comply with federal limits regarding radiofrequency energy deposition and gradient slew rates.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Osorio Suarez, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.